CLINICAL TRIAL: NCT01710605
Title: Randomized Trial to Evaluate the Medico-economic Interest of Taking Into Account Circulating Tumor Cells (CTC) to Determine the Kind of First Line Treatment for Metastatic, Hormone-receptors Positive, Breast Cancers.
Brief Title: Medico-economic Interest of Taking Into Account Circulating Tumor Cells (CTC) to Determine the Kind of First Line Treatment for Metastatic, Hormone-receptors Positive, Breast Cancers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2011-09
Record Dates: First submitted 2012-08-10; First posted 2012-10-19 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Ductal Infiltrating Metastatic Breast Cancer; Hormone-receptors Positive Breast Cancer
Keywords: Circulating tumor cells; Breast Cancer; Hormone-receptors positive
MeSH Terms: conditions — Neoplastic Cells, Circulating; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Active Comparator): Treatment choices (hormonotherapy or chemotherapy) are done according to standard of each center based on clinical, radiological and biological information.
  Interventions: Biological: Circulating tumor cells counting at baseline
- Circulating Tumor Cells (Experimental): Treatment choices (hormonotherapy or chemotherapy) are done according to the number of CTC / 7.5 ml of blood at baseline :
  If <5 CTC : Hormonotherapy If 5 or more CTC : chemotherapy
  Interventions: Biological: Circulating tumor cells counting at baseline

INTERVENTIONS:
Biological: Circulating tumor cells counting at baseline — 20 ml blood sample collected before randomization

SUMMARY:
The STIC CTC study is a randomized trial to evaluate the medico-economic interest of taking into account circulating tumor cells (CTC) to determine the kind of first line treatment for metastatic, hormone-receptors positive, breast cancers. In the standard arm, the kind of treatment will be decided by clinicians, taking into account the criteria usually used in this setting. In the CTC arm, the type of treatment will be decided by CTC count: hormone-therapy if <5CTC/7.5mll (CellSearch technique) or chemotherapy if =5. The main medical objective is to demonstrate the non-inferiority of the CTC-based strategy for the progression-free survival: 994 patients are needed, and will be accrued in French cancer centers. Secondary clinical objectives are to compare toxicity, quality of life and overall survival between the two arms. The medico-economic study will compare cost per progression-free life years gained of the two strategies. The financial impact of centralized (one platform) vs decentralized (several platforms) CTC testing will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women with metastatic ductal adenocarcinoma breast cancer
* 18 years old or more
* Hormone receptors positive breast cancer (ER+ and/or PR+) on the last pathological analysis available.
* Acceptable patient's clinical situation compatible with chemotherapy or hormonotherapy administration
* PS <4
* Life expectancy > 3 months
* Evidence of measurable or evaluable disease (RECIST 1.1 criteria)in the 28 days before selection
* Information of the patient and signature of the informed consent form

Exclusion Criteria:

* Patient treated by chemotherapy or hormonotherapy for their metastatic disease (treatment failure under adjuvant hormonotherapy are accepted)
* Her2 positive breast cancer
* History of other stage II or III cancer in the 5 years. History of other metastatic cancer (whatever the time between the two cancers).
* Persons deprived of their freedom or under guardianship.
* Women unable to comply with the medical follow-up of the study for geographical, social or mental reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2012-02; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival evaluation | 2 years
  According to RECIST 1.1 criteria
Economic evaluation | 2 years
  Economic impact of the strategy will be evaluated (standard treatment choice vs CTC based treatment choice)

SECONDARY OUTCOMES:
Assessing patient quality of life | 2 years
  QLQC30 and BR23 individual questionaries
Evaluation of treatment safety according to NCI-CTCAEv4.03 | 2 years
  Evaluation of both chemotherapy and hormone therapy will be recorded in CRFs whatever the randomization.
Overall survival evaluation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Pierga, Principal Investigator — Institut Curie
Locations (17):
- France (17):
  - Centre François Baclesse, Caen
  - Centre Georges Francois Leclerc, Dijon
  - Clinique Victor Hugo, Le Mans
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Chu Montpellier, Montpellier
  - Institut régional du Cancer de Montpellier, Montpellier
  - Centre Azureen de Cancerologie, Mougins
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Hopital SAINT-LOUIS, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Tenon, Paris
  - Institut Curie - Hopital Rene Huguenin, Saint-Cloud
  - Institut de Cancerologie de L'Ouest - Rene Gauducheau, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Bidard FC, Kiavue N, Jacot W, Bachelot T, Dureau S, Bourgeois H, Goncalves A, Brain E, Ladoire S, Dalenc F, Gligorov J, Teixeira L, Emile G, Ferrero JM, Loirat D, Cabel L, Kadi A, Dieras V, Alix-Panabieres C, Pierga JY. Overall Survival With Circulating Tumor Cell Count-Driven Choice of Therapy in Advanced Breast Cancer: A Randomized Trial. J Clin Oncol. 2024 Feb 1;42(4):383-389. doi: 10.1200/JCO.23.00456. Epub 2023 Nov 6. PMID 37931185
- [Derived] Bidard FC, Jacot W, Kiavue N, Dureau S, Kadi A, Brain E, Bachelot T, Bourgeois H, Goncalves A, Ladoire S, Naman H, Dalenc F, Gligorov J, Espie M, Emile G, Ferrero JM, Loirat D, Frank S, Cabel L, Dieras V, Cayrefourcq L, Simondi C, Berger F, Alix-Panabieres C, Pierga JY. Efficacy of Circulating Tumor Cell Count-Driven vs Clinician-Driven First-line Therapy Choice in Hormone Receptor-Positive, ERBB2-Negative Metastatic Breast Cancer: The STIC CTC Randomized Clinical Trial. JAMA Oncol. 2021 Jan 1;7(1):34-41. doi: 10.1001/jamaoncol.2020.5660. PMID 33151266